CLINICAL TRIAL: NCT03123575
Title: Polypharmacy and Clinically Significant Drug Interactions Among HIV-Infected Patients Receiving Antiretroviral Therapy in The Region Of Madrid: A Population-Based, Cross-Sectional Study
Brief Title: Polypharmacy and Clinically Significant Drug Interactions Among HIV-Infected Patients Receiving Antiretroviral Therapy
Acronym: PODIUM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); SERMAS (Unknown); Molecular-Clinical Pharmacol/Instit.Translational Medicine/University Liverpool (Unknown)
Responsible Party: Sponsor
Other Study IDs: FIBHGM-EONC002-2016
Record Dates: First submitted 2017-04-17; First posted 2017-04-21 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This will be a cross-sectional population-based study carried out in the region of Madrid (6,468,322 inhabitants according to current census) to quantify the number of Co-meds in HIV-infected individuals on ART in the region of Madrid, categorized by age and gender, and to compare the number of Co-meds between the ART-treated population and HIV-uninfected population in the region of Madrid, categorized by age and gender.

DETAILED DESCRIPTION:
This will be a cross-sectional population-based study carried out in the region of Madrid (6,468,322 inhabitants according to current census) to quantify the number of Co-meds in HIV-infected individuals on ART in the region of Madrid, categorized by age and gender, and to compare the number of Co-meds between the ART-treated population and HIV-uninfected population in the region of Madrid, categorized by age and gender.

ELIGIBILITY:
Inclusion Criteria:

* patients who picked-up Co-meds in the study period

Exclusion Criteria:

* NONE

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: ART-treated patients who picked up ARVs and of all HIV-uninfected individuals who picked up Co-meds in the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
the number of Co-meds in HIV-infected individuals on ART | 6 months
  number of Co-meds in HIV-infected individuals on ART in the region of Madrid, categorized by age and gender.
number of Co-meds between the ART-treated population and HIV-uninfected | 6 months
  the number of Co-meds between the ART-treated population and HIV-uninfected population in the region of Madrid, categorized by age and gender.
prevalence of potential CSDIs between ARVs and Co-meds in ART-treated individuals | 6 months
  prevalence of potential CSDIs between ARVs and Co-meds in ART-treated individuals, with description of the types of harm expected from each different potential CSDIs identified

IPD SHARING:
Plan to Share IPD: No